CLINICAL TRIAL: NCT01457742
Title: Non-thermal Pulsed Radio Frequency for Pain Amelioration in Adults With Knee Osteoarthritis: A Double-blind, Randomized, Sham-controlled Trial
Brief Title: Effectiveness Study of the Ivivi SofPulse for Pain Amelioration in Adults With Mild to Moderate Knee Osteoarthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Amp Orthopedics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Ivivi-OAPain-001
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsed Radio Frequency (PRF) (Active Comparator)
  Interventions: Device: Ivivi SofPulse
- Sham (Sham Comparator): Use of Sham device for 15 minutes simulated treatment twice per day
  Interventions: Device: Ivivi SofPulse

INTERVENTIONS:
Device: Ivivi SofPulse — 15 minute Pulsed Radio Frequency (PRF) treatment twice per day
  Arms: Pulsed Radio Frequency (PRF)
Device: Ivivi SofPulse — 15 minute simulated treatment using Sham Device twice per day
  Arms: Sham

SUMMARY:
The purpose of this study is to determine the effectiveness of non-thermal Pulsed Radio Frequency (PRF) treatment with the Ivivi SofPulse for amelioration of knee pain in patients with mild to moderate Osteoarthritis and to determine the duration of clinical benefit following discontinuation of treatment.

DETAILED DESCRIPTION:
This prospective, double-blind, randomized, sham-controlled clinical trial will investigate the effectiveness of PRF using the Ivivi SofPulse on knee pain severity in adults with mild to moderate knee OA. Potential subjects will complete questions related to medical history, inclusion / exclusion criteria, and OA symptom severity. Knee radiographs will be evaluated by the Principal Investigator (PI) or co-investigator for determination of knee OA severity based on the Kellgren/Lawrence criteria. Eligible subjects will enter a 1-week run-in period. After successful completion of the run-in period, subjects will be randomized to PRF treatment twice a day (Active) or sham treatment twice a day (Sham). All subjects will be followed for 4 weeks for purposes of the primary endpoint evaluation. Thereafter, the subjects initially allocated to Active will be equally allocated to Active or Sham and will be followed through 26 or 8 weeks, respectively. The subjects originally assigned to Sham will maintain this treatment regimen through 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 80 years
* Bilateral weight-bearing anteroposterior x-ray of each knee taken within the last 12 months and radiographs submitted to the Principal Investigator for evaluation
* Radiographic evidence of mild to moderate (Kellgren/Lawrence grade 2 or 3) OA in at least one knee based on a weight-bearing anteroposterior x-ray taken within the last 12 months
* Self-reported persistent knee pain severity of 4.0 to 8.0 cm on a 10 cm VAS for most days in the previous 2 months in at least one knee, with grade 2 or 3 OA
* Able to read and complete English-language surveys
* Daily access to the internet
* Ability of the participant to comprehend the full nature and purpose of the study including possible risks and side effects
* Consent to the study and willing to comply with study methods

Exclusion Criteria:

* Subjects who have any implanted metallic leads, wires, or systems (e.g. pacemaker, implantable cardioverterdefibrillator)
* Self-reported persistent knee pain severity > 8.0 cm on a 10 cm VAS in either knee for most days in the previous 2 months
* Radiographic evidence of severe (Kellgren/Lawrence grade 4) OA in either knee based on a weight-bearing anteroposterior x-ray taken within the last 12 months
* Self-reported diagnosis of autoimmune or inflammatory arthritis (e.g. Rheumatoid Arthritis, Lupus, etc.)
* More than 8 days of narcotic pain medication in the last 30 days
* Joint surgery, tidal lavage, or arthroscopy of either knee in the past 6 months
* Intra-articular corticosteroid or hyaluronic acid injections of either knee in the past 6 months
* Oral prednisone use in the past 30 days
* Participation in any clinical trial in the past 30 days
* Knee OA associated with worker's compensation or accident litigation
* Regular use of a walker or wheelchair
* Vulnerable populations including prisoners and nursing home residents
* Anticipated move away from immediate area in next 6 months
* Any medical condition that, in the opinion of the investigator, may compromise patient safety or confound the assessment of treatment effectiveness

After 1-week Run-in Period

* Daily average of "current" knee pain severity < 4.0 cm, assessed on a 10 cm VAS, during the 1-week run-in period in both knees
* Daily average of "current" knee pain severity > 8.0 cm, assessed on a 10 cm VAS, during the 1-week run-in period in either knee
* Daily average of "current" knee pain severity of 4.0 to 8.0 cm, assessed on a 10 cm VAS, during the 1-week run-in period in any knee with Kellgren/Lawrence grades of 0 or 1 in the same knees
* Narcotic use of more than 2 days during the 1-week runin period
* Noncompliance with online symptom reporting requirements

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
A comparison of changes in VAS pain scores at 4 weeks over baseline. | Four weeks
  Comparison of changes in "current" knee pain severity at 4 wks over baseline. Between-group difference of at least 25 percentage points considered clinically significant. "Current" knee pain severity assessed on a 10 cm visual analogue scale, 0 (no pain) and 10 (pain as bad as it can be). The knee that meets radiographic criteria for mild or moderate knee OA and has the highest knee pain severity based on the average daily severity score during the 1-wk run-in period will be selected for the primary endpoint analysis.

SECONDARY OUTCOMES:
Change in knee pain severity and duration of clinical benefit following treatment. | Four weeks
  "Maximum" knee pain severity assessed on a 10 cm VAS and pain improvement
EuroQol EQ-5D | Four weeks
  Improvement of quality of life
OMERACT-OARSI Responder Rate | Four weeks
  Change in need of pain medications and modalities due to knee pain
Adverse events | Four weeks
  Occurance of Adverse Events during treatment period
Treatment compliance | Four weeks
  Improvement of pain and decrease in pain medication with compliant use of the PRF study device as compared to the Sham device.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lane, M.D., Principal Investigator — Mytrus, Inc.
Locations (1):
- Mytrus, Inc., San Francisco, California, United States

REFERENCES:
- See also: website for Mytrus — http://www.mytrus.com